CLINICAL TRIAL: NCT04108962
Title: Phase IV, Single-Center, Open-Label Study Evaluating the Effects of an Anti-IL5 Receptor Alpha (Benralizumab) Monoclonal Antibody in the Treatment of Severe Asthma in Patients With Allergic Bronchopulmonary Aspergillosis
Brief Title: Benralizumab in the Treatment of Patients With Severe Asthma With ABPA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult to find eligible patients willing to participate.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 019-294
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: ABPA; Severe Asthma; Allergic Bronchopulmonary Aspergillosis
Keywords: ABPA; Benralizumab
MeSH Terms: conditions — Asthma; Aspergillosis, Allergic Bronchopulmonary | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Benralizumab treatment will be given by injections administered every 4 weeks for the first 3 injections with an additional injection eight weeks to follow for a total of 16 weeks active treatment
  Interventions: Drug: Fasenra, 30 Mg/mL Subcutaneous Solution

INTERVENTIONS:
Drug: Fasenra, 30 Mg/mL Subcutaneous Solution — Anti-IL5 receptor alpha monoclonal antibody
  Other Names: Benralizumab

SUMMARY:
Phase IV, open-label study will evaluate effects of Benralizumab in the treatment of severe asthma in patients with allergic bronchopulmonary aspergillosis

DETAILED DESCRIPTION:
Subjects who have been identified to have severe asthma with ABPA will be consented and enrolled in the study to receive benralizumab injections administered every 4 weeks for the first 3 injections with an additional injection eight weeks to follow for a total of 16 weeks active treatment with a follow-up/termination visit eight weeks from the last injection. The termination visit will occur week 24 for subjects who complete the study treatment. Subjects who receive the first dose of benralizumab but withdraw from the study or terminate study treatment for any reason should complete all the procedures outlined for the termination visit.

ELIGIBILITY:
SELECT INCLUSION CRITERIA

* Female and Male patients aged 18-75 years inclusively at the time of Visit 1 with a physician diagnosis of Allergic Bronchopulmonary Aspergillosis has met the ISHAM Working Group Diagnostic Criteria for ABPA:

  * Predisposing condition: Bronchial asthma
  * Obligatory criteria (both should be present)

    * Type I aspergillus skin test positive (immediate cutaneous hypersensitivity Aspergillus antigen) or elevated IgE level against Aspergillus fumigatus (Af)
    * Aspergillus niger or Aspergillus flavus may be eligible provided antigen-specific IgE and IgG measurements are available for use.
    * Elevated total IgE levels (>1,000IU/mL)*
  * Other criteria (at least two of three)

    * Presence of precipitating or IgG antibodies against Af in serum
    * Radiographic pulmonary opacities consistent with ABPA
    * Total eosinophil count >500 cells/uL in steroid naïve patients (may be historical)

      * (if the patient meets all other criteria, an IgE value <1,000 IU/mL may be acceptable)
* Severe chronic asthma (for at least 12 months) requiring treatment with high dose ICS plus asthma controller prior to Visit 1

  * Other acceptable asthma controllers include long acting bronchodilators (e.g. a long acting beta-agonist (LABA) or long-acting muscarinic antagonists (LAMA)), a leukotriene inhibitor, theophylline preparations and/or maintenance OCS (daily or every other day OCS requirement in order to maintain asthma control
  * Documented current treatment with high daily doses of ICS ( >500ug of FP equivalent) plus at least one other asthma controller for at least 3 months prior to Visit 1

    * For ICS/LABA combination preparation, highest-strength maintenance doses approved in the U.S. will meet this criterion
    * If the ICS and the other asthma controller therapies are given by separate inhalers, then the patient must be on a high daily ICS dose for 3 months prior to entering the study.
* History of at least 2 asthma exacerbations while on ICS plus another asthma controller (see inclusion criterion 2 for examples) that required treatment with systemic corticosteroids (IM, IV, or oral) in the 12 months prior to Visit 1. For patients receiving oral corticosteroids as a maintenance therapy, an exacerbation is defined as a temporary increase of their maintenance dose for a minimum of 3 days.
* Weight > 40kg

SELECT EXCLUSION CRITERIA

* Clinical important pulmonary disease other than asthma with allergic bronchopulmonary aspergillosis (ie. chronic obstructive pulmonary disease (COPD), cystic fibrosis, sarcoid, and pulmonary fibrosis)
* History of anaphylaxis to any biologic therapy
* Known history of allergy or hypersensitivity reaction to benralizumab or any of its components
* Current smokers or former smokers with a smoking history of > 10 pack years. A former smoker is defined as a patient who quit smoking at least 6 months prior to Visit 1.
* Currently pregnant, breastfeeding, or lactating women
* Concurrent enrollment in another interventional or post-authorization safety study, unless it is observational.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Number of steroid requiring exacerbations | 26 Weeks
  Number of asthma exacerbations requiring the initiation of (or temporary increase in) systemic corticosteroids in severe asthma complicated by ABPA

SECONDARY OUTCOMES:
Patient-Reported Quality of Life as assessed by Saint George Respiratory Questionnaire | 26 Weeks
  The change from baseline score in Saint George Respiratory Questionnaire
Asthma Control as assessed by Asthma Control Questionnaire 6 | 26 Weeks
  The change from baseline score in Asthma Control Questionnaire 6
Lung Function (FEV1) | 26 Weeks
  The FEV1 change from baseline to End of Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Mageto, MD, Principal Investigator — Baylor Scott and White Health
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
no subjects enrolled

REFERENCES:
- [Derived] Kao CC, Hanania NA, Parulekar AD. The impact of fungal allergic sensitization on asthma. Curr Opin Pulm Med. 2021 Jan;27(1):3-8. doi: 10.1097/MCP.0000000000000740. PMID 33027187